CLINICAL TRIAL: NCT05971966
Title: Effect of Virtual Reality Rehabilitation and Muscle Energy Technique in Patients With Patellofemoral Pain Syndrome.
Brief Title: Effects of Virtual Reality Rehabilitation and Muscle Energy Technique in Patients With Patellofemoral Pain Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01652 Nayab Mehmood
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Patellofemoral Pain Syndrome; Knee Pain Chronic
Keywords: muscle energy technique; virtual reality technique; knee pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality technique (Active Comparator): Virtual reality technique+ Conventional PT
  Interventions: Other: Virtual Reality technique
- Muscle energy technique (Experimental): Muscle energy technique + Conventional PT
  Interventions: Other: Muscle energy technique

INTERVENTIONS:
Other: Virtual Reality technique — They would be receiving treatment as follow:
  Specific exercises by using virtual reality with conventional treatment. The VR game included holopoint,hot squat and portal stories that will target the hamstring, quadriceps and gluteas muscles.Frequency: 3 times/week for 4 weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: virtual reality gaming exercises Conventional PT including patellar mobilization+ ultrasound on anterior knee in supine lying + stretching of ITB . Frequency: 10 reps with 5 sec hold for 3 times/week for 4 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 mins
  Arms: Virtual Reality technique
Other: Muscle energy technique — They would be receiving treatment as follow:
  Muscle energy technique of quadriceps and hamstring muscles. Frequency: 3 times/week for 4 weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: Muscle energy technique to improve range of motion.
  Conventional PT including patellar mobilization + ultrasound on anterior knee in supine lying + stretching of ITB. Frequency: 10 reps with 5 sec hold for 3 times/week for 2 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 mins
  Arms: Muscle energy technique

SUMMARY:
The aim of this randomized controlled trial is to determine the effects of Virtual reality rehabilitation and muscle energy techniques in patients with patellofemoral pain syndrome for reducing pain, enhancing knee range of motion and improve functional activities.

DETAILED DESCRIPTION:
Muscle energy technique is defined as a manual treatment in which patient produces a contraction in a precisely controlled position and direction against the counterforce applied by a manual therapist. Applications of MET to stretch and increase myofascial tissue extensibility seem to affect viscoelastic and plastic tissue property.

Virtual reality generates a virtual world in three dimensional space through a computer simulation that stimulates user senses, such as sight and hearing, making users feel as if they are immersed in it. VRBR is effective in improving knee pain, ROM, strength and functions. immersive VR is more appropriate for pain reduction, improving range of motion and functional activities. It distracts the patient and allows to perform active and rehabilitation exercises to reduce cognitive attention in pain and avoidance behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-40
* Both males and females
* Retropatellar or anterior knee pain for atleast past 3 months
* Having knee pain in atleast 2 activities among stair ascent and descent,squatting over 90 degrees, running,jumping,kneeling and prolong sitting with knees flexed.
* Experience pain in one of the following knee tests; a) pain on patellar grinding test, b) pain on apprehension test, c) pain during resisted extension of the knee during 90 degree flexion

Exclusion Criteria:

* Cervical radiculopathy
* Neurological disorder
* Pregnancy
* Rheumatoid arthritis
* Hip or ankle injuries
* Patellar instabilities
* Meniscal or ligament tear
* Who have visual or auditory problems
* With cognitive issues
* Previous surgery related to lower limbs/ radiculopathy
* having received knee injections of corticosteroids or hyaluronic acid
* knee osteoarthritis
* drug use that affects the balance during the past 72 h.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Kujala questionnaire | 4 weeks
  It is a self administered questionnaire for patients with PFPS that consists of 13 questions that relate to specified activities, pain severity, and clinical symptoms. The scores range from a maximum of 100 to a minimum of 0, with lower scores indicating greater pain and disability.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 4 weeks
  VAS is a qualitative pain measurement tool that assigns integer numbers between zero and 10 to different pain levels, where zero means no pain and 10 means excruciating pain. VAS is a reliable scale to measure knee pain
Goniometer | 4 weeks
  It is an instrument that measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Kinza Anwar, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Dr.z pain & brain physiotherapy center, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No